CLINICAL TRIAL: NCT04578899
Title: A Prospective Multicenter Randomized Blind Placebo-controlled Trial "The Effectiveness of Transvertebral Magnetic Neuromodulation in Patients With Detrusor Overactivity"
Brief Title: "The Effectiveness of Transvertebral Magnetic Neuromodulation in Patients With Detrusor Overactivity"
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Joint-Stock Company North-West Center for Evidence-Based Medicine, Russian Federation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1/2020
Record Dates: First submitted 2020-09-15; First posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Intervention Model Description: In case of presence/absence of inclusion/exclusion criteria and written informed consent will be obtained, patients will be randomized in a 1:1 ratio according to the list of randomized blocks using a computer generator. Patients will be randomized at the last available moment in order to minimise bias.
Who Masked: Participant
Masking Description: The hidden distribution of patients will be made with using sequentially numbered sealed opaque envelopes containing the patient's digital code. The randomization code will be recorded in the participant's notes, the patient report form. Then the "sent out" code will be provided to the doctor to prepare a stimulation or placebo.Blinding during the study will be achieved by using a specialized "placebo" function built into the magnetic stimulator "Neuro-MS/d Therapeutic". When using this option, the patient will hear the characteristic sound of the device running, but full pulse stimulation will not be performed. Patients will be deprived of information about the treatment received (stimulation/placebo).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transvertebral magnetic stimulation (Experimental group) (Active Comparator): Experimental intervention will receive non-invasive transvertebral magnetic stimulation of the sacral spine roots (level S2-S3).
  Interventions: Device: Transvertebral magnetic stimulation
- Transvertebral magnetic stimulation (Control group) (Placebo Comparator): Control group will receive an equivalent number of "stimulation" sessions using the placebo option.
  Interventions: Device: Transvertebral magnetic stimulation

INTERVENTIONS:
Device: Transvertebral magnetic stimulation — Continuous theta-burst with a frequency of 5 Hz, lasting 20 minutes 3 times a week for 5 weeks, the total number of procedures is 15

SUMMARY:
The main hypothesis of this study is that magnetic neuromodulation can be used to correct bladder overactivity. The investigators assume that the transvertebral magnetic stimulation can improve both the subjective state of patients evaluated through questionnaires and objective parameters evaluated through invasive and non-invasive urodynamic studies. This study will compare two protocols for magnetic stimulation of the sacral spine roots (S2-S3 segments). The investigators propose to find out the dependence of the therapeutic effect on the frequency of stimulation, the frequency of procedures and the duration of the treatment course.

DETAILED DESCRIPTION:
The aim of the study is to test the hypothesis that the use of magnetic stimulation of the sacral spine roots (S2 - S3) in patients with idiopathic overactive bladder (OAB) will help reduce the clinical and urodynamic manifestations of bladder overactivity.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years;
2. Signed informed consent;
3. The presence of OAB symptoms: urinary frequency, nocturia, urgency and urge incontinence;
4. The presence of detrusor overactivity patterns based on the results of the urodynamic study (UDI)

Exclusion Criteria:

1. The patient, who have been implanted devices that control physiological functions (a pacemaker, a device for deep brain stimulation and chronic epidural brain stimulation, a cochlear implant).
2. Convulsive attacks in the anamnesis;
3. Taking medications that may trigger the risk of seizures;
4. Pregnancy or suspicion on it;
5. The presence in the patient's body of metal elements or objects made with the use of ferromagnets (joint prostheses, eye prostheses, tattoos made using metal ink, surgical clips, staples and other metal suture materials, etc.)
6. Chronic cardiovascular and cerebrovascular diseases in the stage of decompensation or recent acute conditions (myocardial infarction, brain stroke, etc.)
7. Pelvic organ prolapse (II-IV stages according to the POP-Q system)
8. The presence of urinary tract infection
9. The presence of tumors of the pelvic organs

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-09-04 (Actual); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Change baseline of micturition episodes per day | 4, 12, 24, 48 weeks
  Patients should document how many times they go to the restroom during the day and at night, as well as the loss of urine in stressful situations (coughing, sneezing, laughter, squatting, weightlifting, walking, running), changing liner or absorbent and episodes of urgency and urgency-incontinence. The journal shall be held for a consecutive period of 24 hours, for a minimum of three consecutive days.

SECONDARY OUTCOMES:
OAB-Q SF Change Score | Baseline, 4, 12, 24, 48 weeks
  Individual participant change score on the Overactive Bladder Questionnaire short-form (OAB-q SF) will be compared between the two cohorts by student's t-test. The OAB-q SF is utilized to assess the impact of OAB symptoms on the patient's life, and has been shown to be responsive to reductions in urinary urgency, frequency and incontinence during transvertebral magnetic neuromodulation therapy. The OAB-q SF questionnaire consists of 19 items divided into a 6-item symptom severity (SS) scale and a 13-item health-related quality of life (HRQL) scale, with both scales ranging from 0 to 100. For the OAB-q SS scale a higher score indicates worse symptom severity while for the OAB-q HRQL scale a higher score indicates better quality of life.
PGI-I Change Score | Baseline, 4, 12, 24, 48 weeks
  Treatment success at 4,12,24,48 weeks after initiation of transvertebral magnetic neuromodulation therapy. Treatment success will be defined as a response of "very much better" or "much better" on the Patient Global Impression of Improvement (PGI-I), which is a single item questionnaire that asks respondents to rate their improvement after undergoing treatment on a 7-point Likert scale ranging from "very much worse" to "very much better." Statistical analysis will be by intention-to-treat for the primary outcome. A chi-square test will be utilized to determine if there is a statistically significant difference between the two cohorts and sensitivity analyses will be performed using logistic regression analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Dmitriy Shkarupa, Phd, Principal Investigator — JOINT-STOCK COMPANY "NORTH-WESTERN CENTRE OF EVIDENCE-BASED MEDICINE
Locations (1):
- Joint-Stock Company "North-Western Centre of Evidence-Based Medicine", Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No